CLINICAL TRIAL: NCT05922163
Title: Blood Transfusion Education Using Blended Virtual Reality and Simulation for Nursing Undergraduate Students: a Randomized Controlled Trial
Brief Title: Blood Transfusion Education Using Blended Virtual Reality and Simulation for Nursing Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VR2022
Record Dates: First submitted 2023-06-18; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Blood Transfusion Complication
Keywords: Blood transfusion; Nursing education; Nursing practice; Simulation; Virtual reality
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receive the usual blood transfusion education (i.e. Zoom lecture) with the developed VR (Virtual Reality) video education.
  Interventions: Device: Evidence-based VR simulation
- Control Group (No Intervention): Receive the usual blood transfusion education (i.e. Zoom lecture) only.

INTERVENTIONS:
Device: Evidence-based VR simulation — Evidence-based VR simulation videos on BTs for nursing students were developed, including 1) animated blood formation physiology and side effects of BT and 2) 360° BT nursing practice.
  Arms: Intervention Group

SUMMARY:
Nurse-administered blood transfusion (BT) is a common form of medical treatment, but nursing students are often excluded from participating in and observing BTs during clinical placements. To address clinical placement limitations, nursing educators have increasingly adopted technology-guided simulation pedagogies, including virtual reality (VR) simulation, for nursing students' clinical skills education.

ELIGIBILITY:
Inclusion Criteria:

* All undergraduate nursing students enrolled in the 'Nursing of Adults' course in a pre-licensure program at a Hong Kong university.

Exclusion Criteria:

* Students who had vision impairment to watch VR videos;
* Students who had neck pain/ injury to move their head, or open wound to wear the VR headset;
* Students who experienced nausea and dizziness when watching VR videos;
* Students who had epileptic symptoms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Blood transfusion knowledge scale (optimised version of the routine blood transfusion knowledge questionnaire [RBTKQ-O]) | 12-week
  A 34-item scale with score ranging from 0 to 34, higher scores indicate higher levels of blood transfusion knowledge.

SECONDARY OUTCOMES:
Student satisfaction and self-confidence scale [SSSC] | 12-week
  A 13-item scale with score ranging from 13 to 65, higher scores in both subscales refer to higher satisfaction levels with the intervention and self-confidence in conducting blood transfusion practice, respectively.
General self-efficacy scale [GSES] | 12-week
  A 10-item scale with score ranging from 10 to 40, higher scores indicate higher levels of self-efficacy regarding blood transfusion practice.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No